CLINICAL TRIAL: NCT02625948
Title: Tranexamic Acid for Acute ICH Growth prEdicted by Spot Sign
Acronym: TRAIGE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Liping Liu, Professor of Neurology and Stroke Center, Beijing Tiantan Hospital, Capital Medical University, Ministry of Science and Technology of the People´s Republic of China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D141100000114002
Record Dates: First submitted 2015-12-07; First posted 2015-12-09 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Intracerebral Hemorrhage; Stroke
Keywords: Intracerebral Hemorrhage; tranexamic acid; spot sign
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tranexamic acid (Active Comparator): tranexamic acid
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): 0.9% NaCl
  Interventions: Drug: Tranexamic Acid
- observation(spot sign -) (No Intervention): regular clinical treatment

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Placebo; tranexamic acid

SUMMARY:
The purpose of this study is to determine if computed tomography angiography can predict which individuals with intracerebral hemorrhage will experience significant growth in the size of the hemorrhage. For individuals who are at high risk for hemorrhage growth, the study will compare the drug Tranexamic acid to placebo to determine the effect and safety of on intracerebral hemorrhage growth

DETAILED DESCRIPTION:
The Tranexamic Acid for Acute ICH Growth prEdicted by Spot Sign (TRAIGE) is a is a multicentre, randomized, placebo-controlled, double-blind, prospective, investigator-led, clinical trial of tranexamic acid within 6 hours of intracerebral hemorrhage in patients with contrast extravasation on CTA, 'the spot sign'. ICH patients within 6 hours of symptom onset, with the spot sign as a biomarker for ongoing hemorrhage, and no contraindications for antifibrinolytic therapy were enrolled in TRAIGE. The patient with a spot sign will be randomized to receive either the active treatment or placebo, the patient with no spot sign will be given regular treatment as observation. The trial is anticipated to complete in 36 months from the first subject recruitment , with 240 subjects recruited. A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study. The trial has been approved by IRB(Institutional Review Board) /EC(Ethics Committee) in Beijing Tiantan hospital, Capital Medical University.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting with an acute spontaneous hypertensive Intracerebral hemorrhage

1. CTA evaluation can be accomplished within 6 hours of symptom onset, with "spot sign" positive in CTA original image
2. Age range from 18 to 79 years
3. Randomization can be finished and treatment can commence within 8 hours of symptom onset
4. Informed consent has been received in accordance to local ethics committee requirements

Exclusion Criteria:

1. ICH known or suspected to be secondary to tumour, vascular malformation, aneurysm or trauma
2. Infratentorial ICH
3. Glasgow coma scale (GCS) total score of <8
4. ICH volume >70 ml
5. Parenchymal hemorrhage with ventricle involved, blood completely fills one lateral ventricle or more than half of both lateral ventricles
6. Contraindication of CTA imaging (e.g. known or suspected iodine allergy or significant renal failure)
7. Any history or current evidence suggestive of venous or arterial thrombotic events within the previous 6 months, including clinical, ECG, laboratory, or imaging findings. Clinically silent chance findings of old ischemia are not considered exclusion.
8. Planned surgery for ICH
9. Pregnancy or within 30 days after delivery, or during lactation
10. Use of heparin, low-molecular weight heparin, or oral anticoagulation within the previous 1 week, with abnormal laboratory values
11. Known allergy to tranexamic acid
12. Prestroke modified mRS score of >2

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
hemorrhage growth | 24±2 hours
  either >33% or >6 ml increase from baseline, adjusted for baseline ICH volume

SECONDARY OUTCOMES:
Major thromboembolic events | 30±4 days
  (1) acute myocardial ischemia; (2) acute cerebral ischemia; and (3) acute pulmonary embolism
Poor clinical outcome | 90±7 days
  The Number of patients that is Death or major disability(mRS 4-6)
short-term outcome | 30±4 days
  The Number of patients that with Modified Rankin Scale (mRS) 0-2 at 30±4 days
Other thromboembolic events | 90±7 days
  Other thromboembolic events，such as venous thrombosis and other peripheral arterial embolism
Death due to any cause | 90±7 days
  Number of patients that is Death due to any cause by 90±7 days

OTHER OUTCOMES:
Absolute ICH growth volume | 24±2 hours
  The absolute ICH growth volume compared with the baseline CT scan
Absolute IVH growth volume | 24±2 hours
  The absolute IVH growth volume compared with the baseline CT scan

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Aviation General Hospital, Beijing, Beijing Municipality
  - Beijing Fangshan District Liangxiang Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Haidian hospital, Beijing, Beijing Municipality
  - Beijing Huairou District Hospital, Beijing, Beijing Municipality
  - Beijing Shunyi Hospital, Beijing, Beijing Municipality
  - Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Kailuan general hospital, Tangshan, Hebei
  - Tangshan gongren hospital, Tangshan, Hebei
  - Tangshan people's hospital, Tangshan, Hebei

REFERENCES:
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112
- [Derived] Fu F, Sun S, Liu L, Gu H, Su Y, Li Y. Iodine Sign as a Novel Predictor of Hematoma Expansion and Poor Outcomes in Primary Intracerebral Hemorrhage Patients. Stroke. 2018 Sep;49(9):2074-2080. doi: 10.1161/STROKEAHA.118.022017. PMID 30354984